CLINICAL TRIAL: NCT06658743
Title: Designing Team Clinic for Youth With Type 2 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, lily chao, Principal Investigator, Children's Hospital Los Angeles
Other Study IDs: CHLA-24-00160
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
Keywords: youth onset type 2 diabetes; shared medical appointments; group appointments; pediatric type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents and Young Adult Advisory Council: Youth with type 2 diabetes between the ages of 12 to 18.
- Care Giver Advisory Council: Care givers of youth with Type 2 diabetes.
- Curriculum Reviewers: Multidisciplinary team members (including dieticians, clinicians, social workers, and nurses) that take care of patients with type 2 diabetes.

SUMMARY:
The goal of this study is to learn about if shared medical appointment is an acceptable way to deliver care to youth with type 2 diabetes.

The main question[s] it aims to answer are:

* Design four group activities centered around nutrition therapy, peer interactions, exercise and stress management.
* Design the clinical workflow for implementation phase.

Participants will attend quarterly clinic appointments and group activities and take surveys. Researchers will compare this intervention to standard of care.

ELIGIBILITY:
AYA Advisory Council Inclusion Criteria

* Age 12 to 18 at time of study enrollment
* Receives care for type 2 diabetes
* Willingness to attend all meetings
* English-speaking

Exclusion Criteria • Non-verbal or unable to participate in group activities and discussions

Caregiver Advisory Council Inclusion Criteria

* Age 18 or above
* Caregiver of AYA with type 2 diabetes
* Willingness to attend all meetings
* English- or Spanish-speaking

Exclusion Criteria

* Non-verbal or unable to participate in group activities and discussions

Stakeholder Advisory Board Inclusion Criteria

* Age 18 or above
* On staff at CHLA or UCSF
* Clinical or administrative member of the diabetes clinic
* Willingness to participate in monthly meetings. If unable to attend, willingness to review meeting minutes.

Exclusion Criteria • None

Curriculum Reviewers Inclusion Criteria

* Age 18 or above
* CDCESs, nurses, nurse practitioners, dieticians, social workers or physicians in the diabetes clinic
* Clinical members of the diabetes clinic

Exclusion Criteria

• Member of the Stakeholder Advisory Board

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: AYA Advisory Council: Participants will include AYAT2D between the ages of 12 to 18.
  Caregiver Advisory Group: Participants will include caregivers of AYAT2D.
  The Stakeholder Advisory Board will include the PI, co-I's, study coordinator, group facilitators (including Certified Diabetes Care and Education Specialists [CDCES], RD, and behavioral health specialist [BH: psychologist and social worker]), clinicians, and clinic administrator.
  The Curriculum Reviewers will include CDCESs, nurses, nurse practitioners, dieticians, social workers or physicians in the diabetes clinic.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Design four group activities for Team Clinic for youth with type 2 diabetes | Baseline to 5 months
  Activities will be prepared for the focus group for the following topics 1. Nutrition Therapy, 2. Peer Interactions, 3. Exercise, 4. Stress Management.
Design Team Clinic for youth with type 2 diabetes workflow | Baseline to 1 year
  Team Clinic in a multidisciplinary care model that includes 1) individual encounter with clinician, 2) group activity, 3) caregiver group discussion, 4) option to consult with nurse, dietician, and/or behavioral health specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Lily Chao, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF, San Francisco, California

IPD SHARING:
Plan to Share IPD: No